CLINICAL TRIAL: NCT05544279
Title: The Effect of Education Given to the Mothers of Children With Hydrocephalus on Caregiver Burden and Anxiety
Brief Title: Caregiver Burden and Anxiety in Mothers of Children With Hydrocephalus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Dilara Keklik, Research Assistant, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 99
Record Dates: First submitted 2022-09-09; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Hydrocephalus
Keywords: hydrocephalus; children; caregiver burden; anxiety
MeSH Terms: conditions — Hydrocephalus; Caregiver Burden; Anxiety Disorders | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: There are 2 groups: experimental and control groups.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group that given education (Experimental): 7 interviews are held. 3 meaurements are explored. In the first measurement (first interview) "Personal information form", Zarit Burden Interview (ZBI), STAI-S and STAI-T are filled in preoperatively within 24-48 hours, and the planned training and booklet are given. Second measurement (4th interview) is done on the phone within the 1st week after discharge. Third measurement (7th interview) is explored within the 4th week after discharge. In the interim interviews, the training is repeated and the questions about the places that were not understood are answered.
  Interventions: Behavioral: Education
- Control group (No Intervention): 1. Interview (pre-test): 1st interview: Personal information form, ZBI, STAI were filled in preoperatively within 24-48 hours. They receive routine care at the hospital 2nd interview (on the phone within the 1st week after discharge): ZBYÖ, STAI-S and Education follow-up form are filled.
  3rd interview (post-test): ZBYÖ, STAI-S and Education follow-up forms were filled on the phone within the 4th week after discharge. A pdf format of the training material was sent to the mothers in the control group via whatsapp application.

INTERVENTIONS:
Behavioral: Education — Education is given about the focused disease and its nursing care management
  Arms: Intervention group that given education

SUMMARY:
This study is being conducted in randomized controlled trial design to determine the effect of the education given to the mothers of children with hydrocephalus on caregiver burden and anxiety levels.

DETAILED DESCRIPTION:
The number of samples to be taken was calculated as a result of the analysis of the scale mean scores in the control group data obtained in the pre-application. At the end of the 3rd measurement, under the assumption that there will be a 20% more decrease in the intervention group compared to the control group, and using the values obtained from the pilot study, it was determined that 20 patients should be included in the experimental and control groups at 5% error, 80% power.

Research eligibility criteria were as follows;

1. Having children with hydrocephalus aged 0-1 years
2. Having a child with a ventriculoperitoneal shunt operation indication,
3. Having a child in the preoperative period
4. Being the primary caregiver of the child
5. Being literate
6. Not having another relative with chronical disease to care for
7. Residing in Adana province
8. Mothers who were open to communication and cooperation were included in the study.

The hypotheses of the study are as follows;

H0: Between the mothers in the control group and the treatment group; H0-1: There is no difference between the groups in terms of Zarit Burden Interview total mean scores.

H0-2: There is no difference between the groups in terms of State Anxiety Inventory total mean scores.

H03: There is no difference between the groups in terms of Trait Anxiety Inventory total mean scores.

H04: There is no relationship between the groups in terms of Zarit Burden Interview and State Anxiety Inventory total mean scores.

H05: There is no relationship between the groups in terms of Zarit Burden Interview and Trait Anxiety Inventory total mean scores.

Before collecting the data, approvals from the Ethics Board (15 May,2020;99) and from the instituations where the study to be conducted were gained. Besides, principles namely "Informed Consent," "Confidentiality and Protection of Confidentiality," and "Respect to Autonomy" principles were fulfilled by explaining the aim of the study to the participants, by reporting that the information obtained would be kept confidential, and by including the individuals who voluntarily wanted to participate in the study.

Zarit Burden Interview, State-Trait Anxiety Inventory and Personal Information Form and Patient Follow-up Form are being used for collecting data. Totally, it was planned to make 7 interviews with the experimental group and 3 interviews with the control group and 3 measurements are made in the experimental and control groups.

Data is being collected with the first interview face-to-face and the last interview with the telephone interview technique. Training booklet was assessed by 5 lecturers in the field of Child Health and Diseases Nursing according to a kind of DISCERN measuring instrument- The Suitability of Written Materials Form. As a result of the analysis, the total score obtained from The Suitability of Written Materials Form was found to be 26.2±1.09, which indicates that the readability rate of the training content is also high. Furthermore, as a result of the evaluation of five experts in the field, necessary changes were made in the training material.

Training about the content in the booklet and the booklet were given to the experimental group in the first meeting. Each training takes about 45 minutes. Booklets in pdf formats are sent to the control group via whatsApp after the interviews were completed.

The content of the training material is topics related to hydracephalus such as what hydrocephalus is, symptoms of hydrocephalus, treatment of hydrocephalus, what shunt is, signs of infection, nutrition and what to do to prevent complications.

ELIGIBILITY:
Inclusion Criteria: 1. Having children aged 0-1 with hydrocephalus 2. Having a child with a ventriculoperitoneal shunt operation indication, 3. Having a child in the preoperative period 4. Being the primary caregiver of the child 5. Being literate 6. Having no other dependents with chronic diseases at home 7. Residing in Adana province 8. Mothers who were open to communication and cooperation were included in the study.

-

Exclusion Criteria:

1. Not having 0-1 year old child with hydrocephalus
2. No child in the preoperative period
3. Those who do not undertake the primary care of the child
4. illiterate
5. Having no other dependents with chronic diseases at home
6. Those who do not reside in Adana
7. Not open to communication and cooperation
8. Mothers with hearing and speech disabilities were excluded from the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — It is aimed to assess the caregiver burden of mothers, therefore just female are included.
Enrollment: 40 (Estimated)
Dates: Start 2020-07-17 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Zarit Burden Interview | through study completion,1 month
  The scale, which is used to evaluate the caregiving difficulties experienced by caregivers of individuals in need of care, was developed by Zarit, Reever, and Bach-Peterson (1980) in 1980. The Turkish validity and reliability study of the scale was carried out by İnci and Erdem (2006).
State-Trait Anxiety Inventory (STAI) | through study completion, 1 month
  Spielberger et al. developed it in 1970 and the validity and reliability study of this scale was carried out by Öner and Le Compte in 1977.
Patient Follow-up form | through study completion, 1 month
  The training follow-up form, which was created by the researcher as a result of the literature review, was filled in twice in the 1st week and 1st month after the first interview. The purpose of this form; To determine the educational issues that the mother needs after discharge and to follow up the shunt complications.

CONTACTS AND LOCATIONS:
Overall Officials: Ayda Çelebioğlu, PhD, RN, Study Chair — Mersin University
Locations (1):
- Çukurova University Balcalı Hospital Health Education and Research Center, Adana, Sarıçam, Turkey (Türkiye)